CLINICAL TRIAL: NCT06957392
Title: Mechanisms and Interventions of Social Reward Modulating Cognitive Control in Internet Gaming Disorder Via the dACC-DLPFC Circuit
Brief Title: Mechanisms and Interventions of Social Reward on Cognitive Control in Internet Gaming Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Collaborators: Bengbu Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dlJiao-035
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Internet Gaming Disorder
Keywords: Internet gaming disorder; Cognitive control; dACC-DLPFC; Social reward
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Systematic self-help training program for enhancing social reward (Experimental): 1. A single-blind randomized controlled trial is conducted. 30 people, assigned to SRI group (Social Reward Intervention group) , will be received a psychological self-help program aimed at enhancing social reward sensitivity.
  2. Assessments including standardized scales, behavioral tests, and neuroimaging are conducted once before and once after the intervention.
  3. During the course, participants will receive twice-weekly online guidance sessions totaling eight sessions, which mainly focus on practicing ACT (Acceptance and Commitment Therapy) psychological skills, checking progress in social reward learning, and monitoring course advancement. Additionally, one to two offline group discussions are held regularly to enhance treatment adherence and ensure active participation in the self-help program.
  4. The entire intervention lasts approximately one month, with follow-up assessments conducted at 3, 6, and 12 months post-intervention.
  Interventions: Behavioral: Systematic self-help training program for enhancing social reward
- general knowledge about Internet Gaming Disorder . (Other): 1. A single-blind randomized controlled trial is conducted. 30 people, assigned to Control group, was provided with standard educational courses introducing general knowledge about Internet Gaming Disorder, while the others are assigned to SRI group (Social Reward Intervention group). Both groups have equivalent learning durations and delivery formats.
  2. Assessments including standardized scales, behavioral tests, and neuroimaging are conducted once before and once after the intervention.
  3. During the course, participants will receive twice-weekly online guidance sessions totaling eight sessions.
  4. The entire intervention lasts approximately one month, with follow-up assessments conducted at 3, 6, and 12 months post-intervention.
  Interventions: Behavioral: general knowledge about Internet Gaming Disorder .

INTERVENTIONS:
Behavioral: Systematic self-help training program for enhancing social reward — Based on previous research, this study has made significant innovations and optimizations within the traditional framework of Acceptance and Commitment Therapy (ACT). We have specifically developed a systematic self-help training module aimed at enhancing social reward, which includes components such as social scenario experience, social skills training, and the improvement of social reward sensitivity.
  A single-blind randomized controlled trial will be conducted, dividing IGD participants into two groups. The SRI group (Social Reward Intervention group) will receive a psychological self-help training program designed to improve social reward, while the other (Control group) will receive a course introducing general knowledge about Internet Gaming Disorder. Both groups will have identical learning durations and modalities. The self-help training consists of 8 sessions, delivered twice weekly through a blended online and offline learning format, lasting approximately one month.
  Arms: Systematic self-help training program for enhancing social reward
Behavioral: general knowledge about Internet Gaming Disorder . — A single-blind randomized controlled trial is conducted. 30 people, assigned to Control group, was provided with standard educational courses introducing general knowledge about Internet Gaming Disorder. Assessments including standardized scales, behavioral tests, and neuroimaging are conducted once before and once after the intervention.
  During the course, participants will receive twice-weekly online guidance sessions totaling eight sessions. The entire intervention lasts approximately one month, with follow-up assessments conducted at 3, 6, and 12 months post-intervention.
  Arms: general knowledge about Internet Gaming Disorder .

SUMMARY:
Internet Gaming Disorder (IGD) involves impaired cognitive control linked to reduced social reward and dACC-DLPFC brain circuit dysfunction. Enhancing social reward may restore this circuit and improve symptoms. This study uses psychological interventions and neuroimaging to explore and treat IGD.

DETAILED DESCRIPTION:
Cognitive control decline is a key factor in the long-term persistence of Internet Gaming Disorder (IGD). The dorsal anterior cingulate cortex (dACC)-dorsolateral prefrontal cortex (DLPFC) circuit serves as the neural mechanism underlying the maintenance of normal cognitive control function. Social reward activities have been shown to enhance the function of both the dACC and DLPFC. IGD patients exhibit reduced social reward sensitivity alongside diminished functional activity in these two brain regions. Our previous research found that psychological interventions aimed at improving cognitive control can alleviate IGD symptoms; however, individuals with poor social interaction still show limited improvement. Based on these findings, we propose the hypothesis that reduced social reward sensitivity in IGD leads to weakened functional connectivity of the dACC-DLPFC circuit, resulting in cognitive control deficits and exacerbation of IGD behaviors. Enhancing social reward is expected to promote functional connectivity within the dACC-DLPFC circuit, thereby improving cognitive control and mitigating IGD symptoms. To test this hypothesis, we will conduct the following studies: (1) Employing a combination of E-Prime behavioral paradigms, event-related potentials (ERP), and neuroimaging techniques to investigate the attenuated facilitative effects of social reward on cognitive control in IGD patients, and examine its correlation with reduced functional connectivity in the dACC-DLPFC circuit. (2) Designing a psychological intervention aimed at enhancing social reward sensitivity, to evaluate its efficacy in improving cognitive control and reducing IGD severity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 35 years, irrespective of gender, having completed a minimum of 9 years of education and capable of effectively cooperating in questionnaire evaluations.
* Consent to actively cooperate in the completion of subsequent follow-up assessments.
* All are right-handed
* The Gaming Disorder Screening (GDSS) Scale score ≥ 47 points;
* The main game played is Honor of Kings; Average weekly gaming time (Honor of Kings) greater than 21 hours, maintained for over one year; More than 50% of daily internet time spent playing online games;

Exclusion Criteria:

* Severe cognitive functional impairments manifested through a history of head trauma, cerebrovascular diseases, epilepsy, etc., or usage of cognitive enhancement drugs in the past 6 months; an intellectual disability with an IQ score less than 70.
* A diagnosis of schizophrenia or other severe mental illnesses as per the DSM-5 criteria.
* Abuse or dependence on other psychoactive substances (excluding nicotine) within the past 5 years.
* Severe organic diseases that might compromise study participation.
* Color blindness or color weakness

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Severity of Gaming Disorder | through study completion, an average of 1 month
  The severity of gaming disorder was assessed using the Gaming Disorder Screening Scale (GDSS), which consists of 18 Likert-scale items. Each item has four response options (1 = never; 2 = sometimes; 3 = often; 4 = always), with a total score range of 18 to 72. Based on receiver operating characteristic (ROC) analysis using ICD-11 as the gold standard, a total score of ≥47 indicates a high risk of gaming disorder
Social Reward | through study completion, an average of 1 month
  Social reward function was measured using the Social Pleasure subscale of the Multidimensional Anhedonia Scale. This subscale includes 4 items, and participants were first asked to list two current or past social activities that brought them happiness, then to respond to each item assessing aspects such as willingness to engage in these activities and the pleasure experienced during participation.
Executive Function | through study completion, an average of 1 month
  Executive function was evaluated using the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A), comprising 75 items scored on a 3-point Likert scale ranging from "never" to "often." Higher scores on the Global Executive Composite (GEC) reflect greater executive function impairment.

SECONDARY OUTCOMES:
Changes of Behavioral Indicators | through study completion, an average of 1 month
  Behavioral measures included performance indices from the Social Incentive Delay Task and a Social Reward-modified Stop-Signal Task, including hit rate, reaction time for correct hits, Stop-Signal Delay (SSD), and Stop-Signal Reaction Time (SSRT). A reduced hit rate and prolonged reaction time under social reward cue conditions in the Social Incentive Delay Task indicate impaired social reward processing. In the Stop-Signal Task, a higher SSD and shorter SSRT under reward conditions compared to no-reward groups suggest that social reward enhances cognitive control.
Changes of Electrophysiological Indicators | through study completion, an average of 1 month
  Event-related potential (ERP) components N200 and P300 elicited during the Stop-Signal Task were analyzed with respect to amplitude and latency. N200 amplitude indexed conflict monitoring, while P300 latency reflected inhibitory control capacity.
Neuroimaging Indicators | through study completion, an average of 1 month
  Functional magnetic resonance imaging (fMRI) was used to assess the strength of functional connectivity between the dorsal anterior cingulate cortex (dACC) and the dorsolateral prefrontal cortex (DLPFC)

CONTACTS AND LOCATIONS:
Overall Officials: Dongliang Jiao, doctor, Study Chair — School of Mental Health, Bengbu Medical University
Locations (1):
- Bengbu Medical University, Bengbu, China

IPD SHARING:
Plan to Share IPD: No